CLINICAL TRIAL: NCT00437411
Title: Healing Through Affective Self-Awareness in Fibromyalgia: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike Hsu (Other)
Collaborators: St. John Providence Hospital (Unknown); Blue Care Network of Michigan (Other)
Responsible Party: Sponsor-Investigator, Mike Hsu, Research Fellow, Clinical Lecturer, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UM-HUM00008669
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2016-10-24 (Estimated); Status verified 2016-10

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Affect; Pain; Fatigue; Sleep; Stress; Quality of Life; Stress, Psychological; Psychophysiology; Randomized Controlled Trials
MeSH Terms: conditions — Fibromyalgia; Pain; Fatigue; Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Workshop (Experimental): Affective Self Awareness intervention
  Interventions: Behavioral: Affective Self-Awareness workshop
- Control (No Intervention): Waiting-list control.

INTERVENTIONS:
Behavioral: Affective Self-Awareness workshop — Affective Self Awareness intervention: 90 minute face-to-face consultation with the treating physician, then three 2-hour weekly small-group workshops involving education regarding Mind-Body connections, written emotional expression, meditation, and self-affirmation practices.
  Arms: Workshop

SUMMARY:
The investigators are studying whether a brief three-session mind-body workshop helps people with fibromyalgia. The investigators hypothesize that this workshop will significantly improve pain and other symptoms, compared to usual care.

DETAILED DESCRIPTION:
The affective self-awareness approach presumes that many chronic pain states, such as fibromyalgia (FM), can be effectively treated by encouraging self-awareness of emotional tension. While anecdotally effective in selected patients, this approach has thus far not been tested in a randomized controlled trial. Our purpose is to determine whether an affective self-awareness approach significantly improves pain, tenderness, and other FM symptoms in a random sample of FM patients; and to determine what psychosocial factors predict a favorable response.

Comparisons: changes in ratings of pain, tenderness, and other symptoms between two arms of the study:

* three weekly 2-hour small-group meetings supplemented with daily writing and meditative exercises to enhance affective self-awareness
* usual care

ELIGIBILITY:
Inclusion Criteria:

* fibromyalgia, as defined by American College of Rheumatology 1990 criteria.
* at least 18 years of age.
* have access to transportation to and from Providence Hospital, Southfield, MI.

Exclusion Criteria:

* co-morbid medical conditions capable of causing a worsening of physical functional status independent of FM, including morbid obesity, autoimmune diseases, cardiopulmonary disorders (e.g. angina, congestive heart failure, COPD, chronic asthma), uncontrolled endocrine or allergic disorders (e.g. thyroid dysfunction, Type I diabetes), pregnancy, and malignancy within the preceding 2 years.
* any present psychiatric disorder involving a history of psychosis (e.g. schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder etc.), post-traumatic stress disorder, current suicide risk or history of suicide attempt, or substance abuse within 2 years. Note: Subjects with mood or anxiety disorders otherwise will not be excluded.
* changes in medication regimen within one month prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-04; Primary Completion 2008-10 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Change in average pain according to the Brief Pain Inventory | 6 months

SECONDARY OUTCOMES:
Change in Multi-dimensional Fatigue Inventory | 6 months
Medical Outcomes Study sleep subscale | 6 months
Perceived Stress Scale | 6 months
SF-36 Physical Functional Status | 6 months
Profile of Mood States | 6 months
Tender point count | 6 months
Dolorimeter tender point score | 6 months
Ascending and Multiple Random Staircase thumbnail sensitivity thresholds | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael C Hsu, MD, Principal Investigator — University of Michigan Chronic Pain and Fatigue Research Center
Locations (1):
- St. John Providence Hospital, Southfield, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsu MC, Schubiner H, Lumley MA, Stracks JS, Clauw DJ, Williams DA. Sustained pain reduction through affective self-awareness in fibromyalgia: a randomized controlled trial. J Gen Intern Med. 2010 Oct;25(10):1064-70. doi: 10.1007/s11606-010-1418-6. Epub 2010 Jun 8. PMID 20532650